CLINICAL TRIAL: NCT00006333
Title: Studies of the Pathogenesis and Natural History of Arthritis and Related Conditions
Brief Title: Study of Arthritis and Related Conditions
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000222; 00-AR-0222
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Pathogenesis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Subjects with known or suspected arthritis: Subjects with known or suspected arthritis will be evaluated longitudinally

SUMMARY:
This research protocol will recruit patients with arthritis and related conditions for the purpose of screening patients for treatment protocols, and evaluating the natural history of arthritis and related conditions. Patients will be evaluated clinically, radiographically and serologically, and standardized data will be uniformly collected on all patients. Additional imaging using sensitive MRI methods will be obtained in some patients. The collected blood and tissue will be utilized for laboratory studies to continue research on the pathogenic mechanisms of rheumatoid arthritis and related autoimmune joint diseases. Data from the history and physical examination as well as several disability questionnaires in the adult and pediatric population will be used to phenotypically characterize these patients and assess outcome and functional status. Any medical care recommended or provided to the patients will be consistent with routine standards of practice and provided in consultation with the patient's referring physician.

DETAILED DESCRIPTION:
This research protocol will recruit patients with arthritis and related conditions for the purpose of screening patients for treatment protocols, and evaluating the natural history of arthritis and related conditions. Patients will be evaluated clinically, radiographically and serologically, and standardized data will be uniformly collected on all patients. Additional imaging using sensitive MRI methods will be obtained in some patients. The collected blood and tissue will be utilized for laboratory studies to continue research on the pathogenic mechanisms of rheumatoid arthritis and related autoimmune joint diseases. Data from the history and physical examination as well as several disability questionnaires in the adult and pediatric population will be used to phenotypically characterize these patients and assess outcome and functional status. Any medical care recommended or provided to the patients will be consistent with routine standards of practice and provided in consultation with the patient's referring physician.

ELIGIBILITY:
* INCLUSION CRITERIA:

No age limits.

History of inflammatory synovitis of at least one or more swollen joints.

Patient's ability and willingness to give informed consent or in the pediatric patients, the parent's willingness to give informed consent and the patient's willingness to assent to the protocol whenever possible.

EXCLUSION CRITERIA:

None if patients fulfill inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with known or suspected arthritis
Sampling Method: Non-Probability Sample
Enrollment: 697 (Actual)
Dates: Start 2000-10-03 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Determine patterns of arthritis | End of the study
  Evaluate natural history and disease trajectories in rheumatoid arthritis

SECONDARY OUTCOMES:
Confirmatory Studies In RA and related diseases | End of the study
  We would like to continue confirmatory studies and test whether serologic disease markers identified early in the course of the disease are indeed markers of disease severity in patients with more established forms of the disease.
Co-culture experiments using synovial tissue and surgical cartilage specimens | End of the study
  The erosive potential of some but not all forms of arthritis is still poorly understood. We propose to resume co-culture experiments using synovial tissue and surgical cartilage specimens to develop a tissue model of bone erosions using the bioreactor
MRI Imaging in RA and related diseases | End of the study
  We would like to use patients from this cohort to develop the analysis of MRI images, including three dimensionally reconstructed images, and test their use in the evaluation of joint damage and impact on early diagnosis and therapeutic decisions.
Collection of DNA in RA and related diseases | End of the study
  Genetic associations need to be tested in large populations of patients with heterogenous diseases. We would like to continue the collection of DNA in a cohort of clinically well-characterized patients to allow for genetic analysis once a critical body of patients has been collected.
Evaluation of early disability in RA and related diseases | End of the study
  Analysis of the degree of early disability resulting from inflammatory arthritis in the early synovitis cohort patients is currently ongoing. We intend to continue work with the rehabilitation department on the analysis of the extent of disability related to the inflammatory conditions and associated factors in the adult and pediatric population.
Assess cytokine profiles | End of the study
  We would like to comprehensively assess cytokine profiles in the serum of patients with pauciarticular, poly-articular and systemic onset JRA and the influence of response to treatment on cytokine changes.
Correlate the cartilage and bone markers of tissue destruction and repair with MRI images | End of the study
  We would further like to correlate the cartilage and bone markers of tissue destruction and repair with the amount of damage seen on MRI in the different patient disease subsets.
Determine the degree of early disability | End of the study
  Very subtle degrees of early disability have been seen in patients with relatively short disease duration. We would like to determine the degree of early disability in JRA patients and correlate measures of disability with the number, joint location and degree of joint damage on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: James D Katz, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-AR-0222.html